CLINICAL TRIAL: NCT04986592
Title: Recurrent Laryngeal Nerve Monitoring for the Assessment of the Vocal Cords in Thyroid Surgery
Brief Title: Predisection Risk Factors for Vocal Cord Palsy After Total Thyroid Surgery
Status: Completed | Type: Observational
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PR AG 129/2014
Record Dates: First submitted 2021-06-16; First posted 2021-08-03 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Recurrent Laryngeal Nerve Palsy; Risk Factors of Vocal Cord Palsy; Neuromonitoring in Thyroid Surgery
MeSH Terms: conditions — Vocal Cord Paralysis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year

SUMMARY:
In patients undergoing total thyroidectomy, intraoperative nerve monitoring according to the International Standards Guideline Statement may detect nerves more susceptible to injury. The aim of our study was to evaluate the independent risk factors of vocal cord palsy, including those related to pre-dissection nerve monitoring values.

Methods: Prospective observational study in 95 consecutive adult patients undergoing elective total thyroidectomy in Spain. A single experienced phonologist performed a videostroboscopy (VS) exam preoperatively and one week after surgery to assess vocal cord mobility. Each surgical procedure was performed with intermittent intraoperative neuromonitoring. Latency and amplitude values were obtained for the vagal and recurrent laryngeal nerves before surgical dissection and compared with the postoperative VS exam.

DETAILED DESCRIPTION:
After ethics committee approval (PR AG 129/2014), a prospective observational study was carried out at Vall d'Hebron University Hospital, a tertiary hospital in Barcelona, Spain, in accordance with the Standards for Reporting of Diagnostic Accuracy (STARD), including all consecutive adult patients undergoing total thyroidectomy during a 12-month period. All patients understood the various aspects of the study and gave written informed consent. Patient characteristics recorded were age, sex, body mass index, ASA grade, and reason for surgery, among others.

Intraoperative neuromonitoring: Neural monitoring was performed once the carotid neurovascular bundle had been identified and throughout the surgical dissection process to ensure functional integrity of the nerve. We used Avalanche XT® (Dr Langer Medical GmbH, Waldkirch, Germany) equipment fitted with paired electrodes on the tracheal tube, in contact with the vocal cords (7-10 mm above the upper edge of the tube). Intermittent neuromonitoring was performed in each patient according to the international standard guidelines for electrophysiological monitoring20. The VN and RLN were stimulated following the four-step technique (V1: initial vagal stimulation, prior identification and dissection of the VN, R1: initial stimulation of the RLN, R2: post-dissection RLN stimulation, V2: post-dissection vagal stimulation). Vagal stimulation confirmed proper functioning of the entire neuronal circuit, while also avoiding false negatives through stimulation of an injured distal RLN at the lesion site. All signals were recorded on a monitor and collected for evaluation. Vagal and RLN stimulation was programmed at 3 mA and 1 mA, respectively. The event threshold was set to 70-100 uV, and increased to 200 uV, to avoid false-positive events appearing on the monitor due to spontaneous low-level respiratory waves < 100 uV. Electromyographic signals (latency and amplitude) as well as biphasic and triphasic waves were displayed on the monitoring screen. Lack of signal occurred when the monitor showed low-amplitude waves, disturbance of the isoelectric line, multiple waves of variable and scant amplitude, interference or substantial reduction in electromyography response (< 100 uV), and a high-pitched warning sound.

Vocal cords were assessed using VS (Laryngeal Strobe 9400, Pentax Medical, USA) by a single experienced phonologist blinded to the IONM results. The VS exam was performed preoperatively and repeated one week after surgery. The diagnosis of palsy (absence of motion) was made on the basis of an observation of asymmetrical laryngeal motion. Patients with postoperative VCP began voice therapy and were monitored periodically to assess their progress.

Statistics:

The main aim of the present study was to identify independent risk factors for VCP, including those related with pre-dissection IONM values. Continuous variables are expressed as the mean (standard deviation) or the median and interquartile range (i.q.r.) prior to verification of normality by the Kolmogorov-Smirnov test, and categorical variables are expressed as the absolute value (percentage).

The IONM results (response amplitude in uV and latency in ms) were compared with VS findings and classified as true positives (TP) when IONM values were abnormal and VCP was confirmed by VS, as true negatives (TN) when IONM values were normal and vocal cord mobility was normal on VS, as false positives (FP) when IONM values were obviously abnormal but vocal cord mobility was normal on VS, and as false negatives (FN) when IONM values were normal but VS revealed VCP. These IONM results were used to calculate sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV), Youden incidence, with the respective 95% confidence interval (CI).

Perioperative variables included sex, age, BMI, ASA grade, neoplasm diagnosis, lymphadenectomy, and surgery. The bivariate relationship between each factor and the VCP results was analysed using an independent sample t test or the Mann-Whitney U-test, as appropriate, for continuous variables, and using the χ2 or Fisher exact test for dichotomous categorical variables. Receiver operating characteristic (ROC) curves were also plotted to determine the best cut-off points for pre-dissection latency and response amplitude for both VN and RLN to predict postoperative palsy.

These cut-off points were then included in the forward stepwise multivariate logistic regression to identify independent risk factors for VCP. Candidate variables for the logistic regression included sex, age, BMI, neoplasm diagnosis, lymphadenectomy, surgery duration, American Society of Anesthesiologists (ASA) classification, and IONM-related predictive factors such as pre-dissection VN latency, pre-dissection VN response amplitude, pre-dissection RLN latency, and pre-dissection RLN response amplitude.

The odds ratio (OR) and 95% CI were also calculated for all exposure factors. In all cases, the level of significance was set at less than 0.05. The statistical analysis was performed using the software package SPSS version 23.0 (IBM, Armonk, New York, USA).

ELIGIBILITY:
Inclusion Criteria:

* To be at least 18 years old, to accept participation in the study, and to be scheduled for a total bilateral thyroidectomy.

Exclusion Criteria:

* Urgent thyroidectomy, inability to perform videostroboscopy, minor patients, patient refuse to be part of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive adult patients undergoing total thyroidectomy during a 12-month period. All patients understood the various aspects of the study and gave written informed consent.
Sampling Method: Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Response amplitude in recurrent laryngeal nerve in uV | Adult patients undergoing total thyroidectomy during a 12-month period
  Response amplitude reflects summated EMG activity from individual muscle fibers of the thyroarytenoid. We define monitoring waveform response amplitude as the height from the vertical measurement from the apex of the positive waveform deflection to the lowest point in the opposite polarity phase of the waveform ( peak to peak). Lack of signal occurred when the monitor showed low-amplitude response waves, in electromyography response (< 100 uV), and a high-pitched warning sound.
Response amplitude in vagal nerve in uV | Adult patients undergoing total thyroidectomy during a 12-month period
  Response amplitude reflects summated EMG activity from individual muscle fibers of the thyroarytenoid. We define monitoring waveform response amplitude as the height from the vertical measurement from the apex of the positive waveform deflection to the lowest point in the opposite polarity phase of the waveform ( peak to peak). Lack of signal occurred when the monitor showed low-amplitude response waves, in electromyography response (< 100 uV), and a high-pitched warning sound.
Vocal cord palsy | The VS exam was performed one week after surgery, through study completion, an average of 1 yearThe diagnosis of palsy (absence of motion) was made on the basis of an observation of asymmetrical laryngeal motion.
  Vocal cords were assessed using videostroboscopy(Laryngeal Strobe 9400, Pentax Medical, USA) by a single experienced phonologist blinded to the neuromonitoring results

CONTACTS AND LOCATIONS:
Overall Officials: Enric Caubet, Study Director — Hospital Vall d'Hebron , Barcelona. Spain; Marcos De Miguel, Study Chair — Hospital Vall d'Hebron , Barcelona. Spain; Oscar González, Study Director — Hospital Vall d'Hebron , Barcelona. Spain; Mercedes Velasco, Ph, Study Chair — Hospital Universitari Vall d'Hebron Research Institute; Miriam De Nadal, Study Chair — Hospital Vall d'Hebron , Barcelona. Spain; Eva Pelaez, Principal Investigator — Hospital Vall d'Hebron , Barcelona. Spain